CLINICAL TRIAL: NCT03377309
Title: Safety and Tolerability of Perampanel in Amyotrophic Lateral Sclerosis Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study halted due to adverse events
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Johnny Salameh, Associate Professor, American University of Beirut Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM.JS.03
Record Dates: First submitted 2017-12-14; First posted 2017-12-19 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Safety; Tolerability; Perampanel
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — perampanel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fycompa (Experimental): Dose will be increased by 2mg/day increments every one week to reach a maximum dose of 8 mg/day. Treatment phase will be stable dose for 12 weeks then followed by washout period over 2 weeks.
  Interventions: Drug: Fycompa

INTERVENTIONS:
Drug: Fycompa — Dose will be increased by 2mg/day increments every one week to reach a maximum dose of 8 mg/day. Treatment phase will be stable dose for 12 weeks then followed by washout period over 2 weeks.
  Other Names: Perampanel

SUMMARY:
Amyotrophic lateral sclerosis (ALS), the most common motor neuron disease, is a fatal progressive neurodegenerative disease affecting motor cortex, brainstem and spinal cord leading to motor neuron death. It is a devastating disease of the anterior and lateral corticospinal tracts with approximately 3 years mean duration from symptoms onset to death, one-fifth survival at 5 years and only 10% may make it to 10 years.

Among the neuronal death pathways, excitotoxicity mechanism is considered to be the foremost-involved mechanism. AMPA receptors are thought to be the prime mediator of the fast excitation in spinal motor neurons, where they are expressed ubiquitously. AMPA receptor antagonist was able to prevent this acute degeneration in previous animal studies.

The investigators aim to study the tolerability and safety of the novel AMPA antagonist, perampanel, in patients diagnosed with ALS. Perampanel [2-(2-oxo-1-phenyl-5- pyridin-2-yl-1,2-dihydropyridin-3-yl) benzonitrile] with its selective non-competitive AMPA antagonism, was recently approved for epilepsy. Various long-term trials studying perampanel in epilepsy showed favorable tolerability profile and most common side effects were mainly: dizziness, headache and somnolence. All patients presenting to Neurology clinics at AUBMC diagnosed with Amyotrophic Lateral Sclerosis, will be considered for the study. Investigators will obtain informed consents from all patients who agree to be enrolled in this study in accordance with institutional review board (IRB) requirements. Patients of both genders and over 18 years old who meet the El Escorial criteria for possible, probable or definite ALS and fit the inclusion criteria will be recruited. Subjects should not be started on riluzole for the past 30 days or stable on a dose of riluzole for at least 30 days prior to the screening process.

In titration phase, perampanel dose will be increase by 2mg/day increments every one week to reach a maximum dose of 8 mg/day; reaching the maximum dose in four weeks. Treatment phase will be followed by washout period during which, dose will be tapered by 2mg/day every 5 days (over total of 15 days).

ELIGIBILITY:
Inclusion Criteria:

* Amyotrophic Lateral Sclerosis (ALS) volunteers must be diagnosed within the 3 years prior to participation as having possible, probable, or definite ALS, either sporadic or familial according to modified El Escorial criteria
* Age 18-80, able to provide informed consent, and comply with study procedures
* Participants must not have started riluzole for at least 30 days, or be on a stable dose of riluzole for at least 30 days, prior to screening (riluzole-naïve participants are permitted in the study)
* Slow VC test equal to or greater than 50% of the predicted value

Exclusion Criteria:

* The presence of unstable psychiatric disease, cognitive impairment, or dementia that would impair ability of the participant to provide informed consent
* Exposure to any experimental agent within 30 days of entry or at any time during the trial or enrollment in another research study within 30 days of or during this trial
* Women who are breastfeeding, who are pregnant or are planning to become pregnant
* Renal insufficiency as defined by a serum creatinine > 1.5 times the upper limit of normal
* Hepatic insufficiency or abnormal liver function (AST and/or ALT greater than 3 times the upper limit of the normal range)
* Slow VC test less than 50% of the predicted value
* ECG finding of QTc prolongation > 450 ms
* Patients who had already undergone tracheostomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability: Incidence and severity of drug-related adverse effects | During study period up to 4 weeks post- study
  Incidence and severity of drug-related adverse effects

SECONDARY OUTCOMES:
Efficacy: As measured by change in ALSFRS-R score | During study period up to 4 weeks post- study
  Efficacy as measured by change in ALS Functional Rating Scale Revised -ALSFRS-R score ALSFRS-R score is of 12 items with total score of 48(each item score on a scale of 4); 0 reflects severe disability and 48 is the normal score.

CONTACTS AND LOCATIONS:
Overall Officials: Johnny Salameh, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- Johnny S. Salameh, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No